CLINICAL TRIAL: NCT01263678
Title: Helping Patients With Spinal Stenosis Make a Treatment Decision: A Randomized Study Assessing The Benefits of Health Coaching
Acronym: SST HCoach RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22508
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Spinal Stenosis
Keywords: Decisional Conflict; Coaching; Decisional Regret
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Coaching (Other): Usual care for patients with a diagnosis of spinal stenosis after viewing a DA and completing a survey.
  Interventions: Other: Usual Care
- Coaching (Other): Patients randomized to coaching group will receive one week post viewing of Decisional Aid.
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: Coaching — Decision support coaching will be provided after the participant has viewed the decision aid
  Arms: Coaching
Other: Usual Care — Patient views DA and completes post DA survey.
  Arms: Non-Coaching

SUMMARY:
Treatment options for lumbar spinal stenosis include surgical and non-surgical approaches. For most people, the decision depends on how bothered they are by their symptoms and how they feel about having surgery. Since individuals with the same clinical presentation may feel differently about their symptoms and how they view the benefits and harms of their options, there is no agreed upon "best"treatment. It has been shown that, for "preference-sensitive" decisions like this one, decision aids (tools that pair balanced, evidence-based information regarding treatment options with values clarification) improve patients'knowledge and realistic expectations, lower decisional conflict, increase patient involvement in decision making, decrease the number of undecided, and increase agreement between values and choice.1 The Spine Center, in collaboration with the Center for Shared Decision Making (CSDM) at Dartmouth Hitchcock Medical Center (DHMC), has been providing patients with decision aids (DAs) for several years.

Hypothesis:

Patients identified as having low literacy and/or high decisional conflict after viewing a video decision aid will show greater resolution of their decisional conflict, higher decision self-efficacy and less decision regret if a coaching intervention is paired with a video decision aid.

Decision support in the form of coaching develops patients'skills in preparing for a consultation and deliberating about their options.2 A study of women with abnormal uterine bleeding showed that pairing coaching with a DA helped patients clarify their values and preferences, reduced costs, and increased long term satisfaction.3 The investigators plan to assess the impact of coaching in patients with lumbar spinal stenosis who are referred to the CSDM for a video decision aid about their treatment options. The investigators are also interested to learn whether screening for low literacy and high decisional conflict can identify a subgroup of patients who are more likely to benefit from coaching.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Adults over 18

Exclusion Criteria:

* Non-English Speaking
* Anyone under the age of 18
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assess the impact of decision coaching, following a specialty consultation for lumbar spinal stenosis | 1 year
  1. Assess the impact of decision coaching, following a specialty consultation for lumbar spinal stenosis, on levels of decisional conflict.
  2. Assess the impact of decision coaching on decision self-efficacy, the number of treatment decision-related clinical contacts, treatment follow-through and decision regret.
  3. Determine whether we can develop a tool that will allow us to identify patients most likely to benefit from coaching and develop a process to provide coaching to patients who need help making treatment decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Jon D Lurie, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States